CLINICAL TRIAL: NCT00115297
Title: Effects of Montelukast on Early Life Wheezing
Brief Title: Montelukast for Early Life Wheezing
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Craig Lilly, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 192; R01HL080073 (NIH)
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Lung Diseases; Asthma
MeSH Terms: conditions — Lung Diseases; Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Montelukast (Experimental): Participants who are 2 to 3 years old received 5-mg montelukast tablets and participants who are 12 months to 2 years old received 4-mg montelukast granules.
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): Participants who are 2 to 3 years old received 5-mg montelukast placebo tablets and participants who are 12 months to 2 years old received 4-mg montelukast placebo granules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — Participants who are 2 to 3 years old received 5-mg montelukast tablets and participants who are 12 months to 2 years old received 4-mg montelukast granules.
  Arms: Montelukast
Drug: Placebo — Participants who were 2 to 3 years old received placebo montelukast tablets and participants who were 12 months to 2 years old received placebo montelukast granules.
  Arms: Placebo

SUMMARY:
This study will determine the effects of montelukast on the duration of wheezing in children 12 months to 3 years of age who visit a physician for care of a wheezing illness. Only patients from the Ankara area of Hacettepe University Medical Center in Turkey will be included in this study.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma has a large impact on the children of our society. It is among the most common chronic diseases of childhood and is the leading cause of absenteeism from school. It is unknown as to why more children are having recurrent episodes of wheezing and why some children have asthma while others do not. There is increasing evidence that differences in innate immune responses among children can determine which child will have recurrent wheezing and asthma. While many studies have focused on the factors that initiate innate immune responses, there are relatively few studies of the downstream factors that cause abnormal airway responses. There is evidence that eicosanoid mediators are part of the innate immune response and can function as its effector arm for allergic responses. The ability of leukotrienes and prostaglandins to produce central features of the asthma phenotype is well described and there is emerging evidence that lipoxins facilitate restoration of allergic changes in the airways. This study will test the hypothesis that the balance of airway eicosanoid expression during early-life wheezing illness and the genetically determined capacity to respond will predict recurrent wheezing. Moreover, an intervention to restore a more normal tissue response to this imbalance will reduce symptoms of early-life wheezing and subsequent recurrent episodes.

DESIGN NARRATIVE:

This will be a prospective, double-blind, randomized, placebo-controlled, parallel-group study of the effects of montelukast on the duration of wheezing in children 12 months to 3 years of age who are under the care of a physician for a wheezing illness. Study treatment will be given for 56 days. Participants who are 2 to 3 years old will receive either 5-mg montelukast tablets or matching placebo. Participants who are 12 months to 2 years old will receive 4-mg montelukast granules or matching placebo. The primary outcome parameter of this study will be the number of days that the infant is observed to be free of wheezing by the primary caregiver. The secondary outcome parameters will be the number of wheezing episodes during the treatment period and the rate of recurrent wheezing during the follow-up period. The study, which is a consortium arrangement between the Brigham and Women's Hospital and the Hacettepe University Medical Center in Turkey, will recruit children only from the Ankara area of Hacettepe University Medical Center in Turkey.

This study will be one of three, which include: 1) measuring the airway eicosanoid profiles of pediatric "wheezing" patients 3 months to 3 years old; 2) determining if genetic variants in eicosanoid metabolic and response pathways are associated with recurrent wheezing; and 3) determining how intervention with montelukast (singulair) affects symptoms and the rate of recurrent wheezing.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed wheezing illness

Exclusion Criteria:

* Asthma
* Prematurity
* Known intolerance to montelukast

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2004-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig M. Lilly, MD, Study Chair — University of Massachusetts/UMass Memorial
Locations (1):
- University of Massachusetts/UMass Memorial, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from University hospital clinics and inpatient services
Pre-assignment Details: Specialist physician confirmed new onset wheezing and completion of study data gathering instruments.
Groups:
- Monteluksat: 5-mg montelukast tablets or 4 mg granules)
  Montelukast: Participants who are 2 to 3 years old will receive 5-mg montelukast tablets and participants who are 12 months to 2 years old will receive 4-mg montelukast granules.
- Placebo: Placebo (montelukast tablet or montelukast granules)
  Placebo: Participants who are 2 to 3 years old will receive placebo montelukast tablets and participants who are 12 months to 2 years old will receive placebo montelukast granules.
Period: Overall Study
Arm/Group | Monteluksat | Placebo
Started | 30 | 32
Completed | 30 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Montelukast: 5-mg montelukast tablets or 4 mg granules
  Montelukast: Participants who are 2 to 3 years old will receive 5-mg montelukast tablets and participants who are 12 months to 2 years old received 4-mg montelukast granules.
- Placebo: Placebo (placebo tablets or granules)
  Placebo: Participants who are 2 to 3 years old will receive placebo montelukast tablets and participants who are 12 months to 2 years old received placebo montelukast granules.
- Total: Total of all reporting groups
Arm/Group | Montelukast | Placebo | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 13 [8.5 to 19.3] | 11.5 [8.3 to 20.0] | 13.0 [9.0 to 20.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 19 | 21 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 32 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 32 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Wheezing-free Days of Infant (Observed by Primary Caregiver)
Time Frame: First 56 days of study
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Montelukast: 5-mg montelukast tablets
  Montelukast: Participants who are 2 to 3 years old received 5-mg montelukast tablets and participants who were 12 months to 2 years old received 4-mg montelukast granules.
- Placebo: Placebo (montelukast tablets)
  Placebo: Participants who are 2 to 3 years old received placebo montelukast tablets and participants who were 12 months to 2 years old received placebo montelukast granules.
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 30 | 32
Days | 25.5 [10.8 to 37.0] | 30.5 [7.5 to 39.8]

2. Secondary Outcome: Wheezing at Day 7
Time Frame: Study day 7
Measure: Number; unit: participants
Groups:
- Placebo: Placebo (montelukast tablets)
  Placebo: Participants who were 2 to 3 years old received placebo montelukast tablets and participants who were 12 months to 2 years old received placebo montelukast granules.
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 30 | 32
participants | 10 | 22

3. Secondary Outcome: The Number of Participants Requiring Rescue Beta Agonist Use
Time Frame: Measured during the daytime
Measure: Number; unit: participants
Groups:
- Montelukast: 5-mg montelukast tablets or granules
  Montelukast: Participants who are 2 to 3 years old received 5-mg montelukast tablets and participants who were 12 months to 2 years old received 4-mg montelukast granules.
- Placebo: Placebo (tablets or granules)
  Placebo: Participants who were 2 to 3 years old received placebo montelukast tablets and participants who were 12 months to 2 years old received placebo montelukast granules.
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 30 | 32
participants | 15 | 26

ADVERSE EVENTS:
Time Frame: Over the 60 day period of active agent or placebo administration
Groups:
- Montelukast: Montelukast tablets or granules
  Montelukast: Participants who are 2 to 3 years old received 5-mg montelukast tablets and participants who were 12 months to 2 years old received 4-mg montelukast granules.
- Placebo: Placebo (tablets or granules)
  Placebo: Participants who are 2 to 3 years old will receive placebo montelukast tablets and participants who are 12 months to 2 years old will receive placebo montelukast granules.
Arm/Group | Montelukast | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 0/30 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No